CLINICAL TRIAL: NCT01032473
Title: Mechanisms of Sleep Disturbance in Children With Generalized Anxiety Disorder (GAD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's National Research Institute (Other)
Responsible Party: Candice Alfano, Ph.D., Children's National Medical Center
Other Study IDs: CNMC-9978
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Generalized Anxiety Disorder; Sleep Disturbances
MeSH Terms: conditions — Generalized Anxiety Disorder; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary cortisol
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GAD: Children between the ages of 7-11 years diagnosed with Generalized Anxiety Disorder (GAD)
- Control: Children between the ages of 7-11 years free of significant medical or behavioral problems (matched to children diagnosed with GAD based on age, gender, and ethnicity).

SUMMARY:
Anxiety disorders are among the most common mental disorders in children, affecting approximately 1 out of every 10 children and adolescents. Symptoms of anxiety disorders may include excessive fear/anxiety/worry, somatic complaints such as headaches and muscle aches, and impaired social and family relationships. Some children with anxiety also experience sleep problems, however, little is known about the sleep patterns of anxious children. The purpose of the study, conducted at Children's National Medical Center, is to examine the sleep characteristics of children with Generalized Anxiety Disorder (GAD) compared to a control group of children without GAD to see how sleep behaviors and daytime behaviors are related.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common mental disorders in children, affecting approximately 1 out of every 10 children and adolescents. Symptoms of anxiety disorders may include excessive fear/anxiety/worry, somatic complaints such as headaches and muscle aches, and impaired social and family relationships. Some children with anxiety also experience sleep problems, however, little is known about the sleep patterns of anxious children. The purpose of the study, conducted at Children's National Medical Center, is to examine the sleep characteristics of children with Generalized Anxiety Disorder (GAD) compared to a control group of children without GAD to see how sleep behaviors and daytime behaviors are related.

To qualify for this study, participants must first be evaluated via a brief, telephone screening. Qualified families will be invited for a comprehensive diagnostic interview. All parents and children must sign a written consent/assent in order to participate.

Two groups of children are being recruited: children diagnosed with (a primary diagnosis of) GAD and matched, healthy controls. To be included in the GAD group, children must:

* Meet DSM-IV criteria for a primary diagnosis of generalized anxiety disorder (GAD)
* Be between the ages of 7 and 11 years old
* Not take any psychotropic medications
* Not have any chronic/major medical problems
* Be of (at least) average intelligence (i.e., IQ of 80 or greater)
* Not meet criteria for psychosis, bipolar, or major depressive disorder
* Parents and children must be English speaking

To be included in the control group, children must:

* Not meet criteria for a psychiatric or sleep disorder
* Be between the ages of 7 and 11 years old
* Not take any psychotropic medications
* Not have any chronic/major medical problems
* Be of (at least) average intelligence (i.e., IQ of 80 or greater)
* Parents and children must be English speaking

Participation is voluntary. Families who choose to participate will be asked to make two visits to Children's National. During their first visit, children and caregivers will be asked to complete self- and parent-report forms, as well as diagnostic interviews. Children will also be administered an abbreviated intelligence test. During their second visit, which is an optional component of the study, participants (and one parent) will stay overnight at Children's National and children will undergo an overnight sleep (polysomnographic) evaluation. Between these visits, participants will wear wrist actigraphs for seven days. An actigraph is a small device that looks like a watch and measures sleep and wake periods. Families will be called daily during this week-long assessment and administered a brief phone-based assessment regarding children's anxiety symptoms. Participants will receive some compensation for time and travel.

ELIGIBILITY:
Inclusion Criteria:

To be included in the GAD group, children must:

* Meet DSM-IV criteria for a primary diagnosis of generalized anxiety disorder
* Be between the ages of 7 and 11 years old
* Not take any psychotropic medications
* Not have any chronic/major medical problems
* Be of (at least) average intelligence (i.e., IQ of 80 or greater)
* Not meet criteria for psychosis, bipolar, or major depressive disorder
* Parents and children must be English speaking

To be included in the control group, children must:

* Not meet criteria for a psychiatric or sleep disorder
* Be between the ages of 7 and 11 years old
* Not take any psychotropic medications
* Not have any chronic/major medical problems
* Be of (at least) average intelligence (i.e., IQ of 80 or greater)
* Parents and children must be English speaking

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-08

CONTACTS AND LOCATIONS:
Overall Officials: Candice Alfano, Ph.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States